CLINICAL TRIAL: NCT03782974
Title: A Randomized, Placebo-controlled, Triple-blinded Evaluation of Proglucamune® in the Treatment of Protective Qi Deficiency
Brief Title: A Follow-up Trial of Proglucamune® in the Treatment of Protective Qi Deficiency, a TCM Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Collaborators: Elegant And Olive Health Clinic, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201878
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Protective Qi Insufficiency (a Condition Term From TCM)
Keywords: Protective Qi; Immunity
MeSH Terms: interventions — beta-Glucans

STUDY DESIGN:
Intervention Model Description: Individuals with Protective Qi Insufficiency
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, on-site care-providers and investigators, and the outcome assessors will be informed that this study is placebo controlled, and that each participant has a 50/50 chance of receiving treatment or placebo. The test material will include treatment and placebo, both coated by the same coating. The code will be kept by the sponsor and disclosed after the analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proglucamune treatment (Experimental): Participants were treated with 2 tablets of Proglucamune per day (containing 200mg of beta glucan) for a total duration of 8 weeks.
  Interventions: Dietary Supplement: beta glucan
- Placebo (Placebo Comparator): Participants were treated with 2 tablets of placebo per day (contain no beta glucan) for a total duration of 8 weeks.
  Interventions: Dietary Supplement: beta glucan

INTERVENTIONS:
Dietary Supplement: beta glucan — Following screening and enrollment, participants will be treated with 2 tablets (Proglucamune or placebo) per day for a total duration of 8 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).

SUMMARY:
This is a follow-up Phase II study of a previously complete pilot trial (Protocol ID: 201875) with the same goal: evaluating the activity of Proglucamune on Protective Qi (PQi) Insufficiency.

According to Traditional Chinese Medicine (TCM) principle, Protective Qi is a one specific concept of Qi that provides the vital energy of the body. It works primarily on the body surface as a defensive barrier. In this context, Protective Qi is analogous to anatomical barriers of the innate immune system located for example, at the skin surface and the mucosal surfaces of the respiratory and digestive tract. Individuals with PQi Insufficiency are predisposed to frequent cold and other symptoms caused by invasion of external pathogens ("Wai Xie" or "external evil" in TCM).

ß-glucan is a polysaccharide that activates macrophage (Dectin-1) and neutrophil (CR3) receptors, and therefore enhances immune defense at digestive and respiratory mucosa. Clinical trials have shown its immune activity such as preventing upper respiratory tract infection (URTI) and Traveler's diarrhea. Notably, ß-glucan is a component of Ganoderma Lucidum (or Reishi / Lingzhi), one TCM ingredient well-known for improving Qi. Based on this connection, investigators hypothesized that ß-glucan is the active ingredient in Reishi that at least partially accounts for Reishi's activity on Qi.

To test our hypothesis, investigators have conducted an uncontrolled pilot trial that investigated the effect of a commercially available, high ß-glucan containing product, Proglucamune®, on PQi status. Proglucamune contains ß-glucan from three different natural sources: Reishi mushroom, Shiitaki mushroom, and Bakers' yeast, each providing ß-glucan that differs slightly in their molecular structure. The data obtained demonstrated a statistically significant effect of Proglucamune on improving PQi in individuals with PQi Insufficiency. The current study is aimed to further determine this effect in a more stringent (placebo-controlled, randomized, and triple-blinded) way.

DETAILED DESCRIPTION:
Unlike mainstream Western medicine (WM), alternative medicines (AM) such as Traditional Chinese Medicine (TCM), emphasizes individually-differentiated therapies. As such, AM therapies are normally not tested in clinical studies that statistically demonstrate the efficacy at the populational level for applicable patients, and this makes it difficult to objectively evaluate and compare different therapies. The lack of clinical studies stands as a barrier for the advance of AMs as well as their engagement with WM. In fact, most researchers view AMs primarily as untapped sources of "active ingredients/compounds" for drug development, but disregard the rationales under which the therapies were developed. A "One-Way-Traffic" research paradigm is thus created wherein AM therapies are investigated for their efficacy by WM standards, whereas the vast potential of employing WM therapies for AM therapeutics is ignored. In light of this, investigators set up a novel strategy that bridges TCM and WM, i.e., testing a WM-based therapy by TCM standards through clinical trial/statistics- based method.

Qi is a central concept in TCM and was first documented in the oldest TCM writings more than 2000 years ago. Generally speaking, Qi refers to the vital energy of the body and is derived from two primary sources: 1) inborn Qi (that may be construed as genetics), and 2) pectoral Qi (can be construed as metabolism). Moreover, Qi manifests itself in two forms: Nutritive Qi and Protective Qi (PQi), which can be understood to reflect an individual's nutritional state and immune health, respectively. Regarding the latter, protective Qi functions to defend the body from the invasion of external pathogens. TCM also emphasizes that Protective Qi works primarily on the body surface as a defensive barrier. In this context, Protective Qi is analogous to anatomical barriers of the innate immune system located for example, at the skin surface and the mucosal surfaces of the respiratory and digestive tract.

TCM has developed a number of methods to strengthen the Qi. Prominent among these is the use of Reishi, either alone or in combination with other TCM remedies. The use of Reishi was described in detail in the first TCM pharmacopedia "Compendium of Materia Medica" published in year 1,600. Nonetheless, although PQi is part of the general Qi, the specific effect of Reishi on Protective Qi is less documented. Anecdotal reports are available that claim significant improvement of Protective Qi with Reishi or Reishi- containing formulas within days. Notably, WM has identified immune-boosting properties of Reishi, which may explain the Qi enhancing effects of this plant. Specifically, beta-glucan - a component of Reishi - has been shown to activate macrophage (large white blood cells in the immune system that destroy bacteria and other harmful substances), neutrophil (a type of white blood cells that are important for protection against infections), and other immunocytes (cells capable of producing an immune response), and may exhibit particular benefits among macrophage-rich organs such as the lung, liver and spleen. In fact, ß-glucans from sources other than Reishi, such as baker's yeast, are able to initiate the same immune response and clinical benefits.

The overlap of TCM and western medicine concerning the beneficial effects of Reishi for its Qi enhancing and immune-modulating effects, respectively, has prompted us to investigate whether or not Reishi, in conjunction with other natural products used in TCM, can enhance an individual's Protective Qi. A previous Pilot trial has been conducted that aimed to determine if a commercially available dietary supplement (Proglucamune®, USANA Health Sciences) containing powdered Reishi and Shitake mushrooms as well as baker's yeast extract, and which is comprised of 11% ß-glucans by weight, would improve Protective Qi in subjects diagnosed by practitioners of TCM as having low or insufficient Protective Qi. The data obtained demonstrated a statistically significant effect of Proglucamune on improving PQi. Based on the effect size and variability, investigators have arrived, via statistical methods, at the necessary sample size for a more definitive (placebo-controlled, randomized, and triple-blinded) trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females aged 18 to 65 years (inclusive) without regard to race or ethnic background
2. Provide a signed Informed Consent prior to entry in the study.
3. Willing to follow all study instructions and consume the assigned investigational product for 12 weeks.
4. Not currently taking a beta-glucan containing supplement or any other supplement that might interfere with the study design.
5. Ability to swallow tablets and pills.
6. Exhibit an PQi Insufficiency score > 2 (See Primary Outcome Measure)

Exclusion Criteria:

1. Persons diagnosed by TCM as having medical conditions other than low Qi.
2. Significant acute or chronic illness or other medical conditions that will prevent or interfere with giving an informed consent, or with participation in the study.
3. Scheduling difficulties or lack of transportation that will prevent or interfere with their ability to attend all of the necessary study visits.
4. Persons medically diagnosed with depression or anxiety disorders.
5. Persons with a history of alcohol abuse or other substance abuse within the previous 2 years.
6. Females who are attempting to become pregnant, pregnant, lactating or who have given birth within 1 year.
7. Persons who have had a medical surgery in the past 4 weeks or have scheduled a surgery during the study period.
8. Persons currently enrolled in a clinical trial, or who have completed a clinical trial within the last 4 weeks.
9. Allergies to mushrooms or other fungi.
10. Significant problems with constipation or diarrhea.
11. A lifestyle or schedule incompatible with the study protocol.
12. Persons who are allergic to yeast products, have autoimmune disease/an immune disorder, or take antidepressants, blood thinners (anticoagulants, acetylsalicylic acid), or immunosuppressant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 207 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Bernstein, MD, Principal Investigator — Department of Family and Community Medicine, Humber River Hospital
Locations (1):
- Elegant And Olive Health Clinic, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller SD, Yang M, Treadwell MJ, Werner EM, Hassell KL. Patient reports of health outcome for adults living with sickle cell disease: development and testing of the ASCQ-Me item banks. Health Qual Life Outcomes. 2014 Aug 22;12:125. doi: 10.1186/s12955-014-0125-0. PMID 25146160
- [Background] Hays RD, Spritzer KL, Thompson WW, Cella D. U.S. General Population Estimate for "Excellent" to "Poor" Self-Rated Health Item. J Gen Intern Med. 2015 Oct;30(10):1511-6. doi: 10.1007/s11606-015-3290-x. Epub 2015 Apr 2. PMID 25832617
- [Derived] Wu JR, Cheng HJ, Shi JP, Yin WD, Wang J, Ou XQ, Chen JL, Bernstein I, Levy M, Maddela R, Sinnott R, Tian JQ. beta -Glucan Improves Protective Qi Status in Adults with Protective Qi Deficiency-A Randomized, Placebo-Controlled, and Double-Blinded Trial. Chin J Integr Med. 2022 May;28(5):394-402. doi: 10.1007/s11655-021-3444-0. Epub 2021 May 8. PMID 33963479
- See also: description for Global Health Questionnaire (PROMIS® Scale v1.2.) — http://www.healthmeasures.net/explore-measurement-systems/promis
- See also: description for Emotional & Behavioral Dyscontrol Questionnaire (Neuro-QoL) — http://www.healthmeasures.net/explore-measurement-systems/neuro-qol

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 207 enrolled participants, 138 met inclusion criteria and were randomized to treatment.
Groups:
- Proglucamune Treatment: Participants were treated with 2 tablets of Proglucamune per day (containing 200mg of beta glucan) for a total duration of 12 weeks.
  beta glucan: Following screening and enrollment, participants will be treated with 2 tablets (Proglucamune or placebo) per day for a total duration of 12 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).
- Placebo: Participants were treated with 2 tablets of placebo per day (contain no beta glucan) for a total duration of 12 weeks.
  beta glucan: Following screening and enrollment, participants will be treated with 2 tablets (Proglucamune or placebo) per day for a total duration of 12 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).
Period: Overall Study
Arm/Group | Proglucamune Treatment | Placebo
Started | 70 | 68
Completed | 62 | 61
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proglucamune Treatment | Placebo | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.00 [38.25 to 56.00] | 51.00 [44.75 to 57.00] | 50.05 [39.25 to 56.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 109
  Male | 13 | 16 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 68 | 66 | 134
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Protective Qi Deficiency (PQD) [Count of Participants; unit: Participants] — Protective Qi Deficiency of each participant is diagnosed by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  Participants | 60 | 55 | 115
Severity Score of PQD [Mean (Standard Deviation); unit: units on a scale] — The severity score is based upon the weighted diagnosis of 7 symptoms by Traditional Chinese Medicine practitioners. The severity score ranges fronm 1- 5; 5 is considered the worst outcome and the individual exhibits severe PQD; conversely, 1 indicates that the individual exhibits no PQD. The weighted score of the 7 symptoms is: [cold frequency*0.375+ (aversion to wind&cold +spontaneous sweating)/2 +(Pulse*0.3+Cun Pulse*0.5+Tongue*0.25+Low voice*0.2)]/3.
  units on a scale | 2.66 (0.45) | 2.58 (0.36) | 2.62 (0.41)
Tongue [Median (Inter-Quartile Range); unit: units on a scale] — The range of the tongue score is 1- 5 and 5 is considered the worst outcome. It is scored by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  units on a scale | 3.50 [3.00 to 4.00] | 3.50 [3.00 to 4.00] | 3.50 [3.00 to 4.00]
Low voice & apathy [Median (Inter-Quartile Range); unit: units on a scale] — The range of the Low voice & apathy(II) score is 1- 5 and 5 is considered the worst outcome. It is scored by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  units on a scale | 3.00 [2.50 to 3.00] | 2.50 [2.00 to 3.00] | 2.50 [2.00 to 3.00]
Cold frequency [Count of Participants; unit: Participants] — It is a standardized numerical interval scale. The range of it is 0 - 3, and 3 is the worst outcome
  Score 0: No cold in the past 2 months
  Score 1: Once in the past 2 months
  Score 2: Twice in the past 2 months
  Score 3: 3 times or more in the past 2 months
  Participants
    None | 17 | 14 | 31
    Once | 42 | 44 | 86
    Twice | 10 | 10 | 20
    Three Times | 1 | 0 | 1
Spontaneous sweating [Median (Inter-Quartile Range); unit: units on a scale] — The range of the Spontaneous Sweating score is 1- 5 and 5 is considered the worst outcome. It is scored by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  units on a scale | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00]
Aversion to wind & cold [Median (Inter-Quartile Range); unit: units on a scale] — The range of the Aversion to wind & cold score is 1- 5 and 5 is considered the worst outcome. It is scored by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  units on a scale | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00]
Overall Pulse [Median (Inter-Quartile Range); unit: units on a scale] — The range of the Overall Pulse score is 1- 5 and 5 is considered the worst outcome. It is scored by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  units on a scale | 3.50 [3.00 to 4.50] | 3.50 [3.00 to 3.80] | 3.50 [3.00 to 4.00]
Cun Pulse [Mean (Standard Deviation); unit: units on a scale] — The range of the Cun Pulse score is 1- 5 and 5 is considered the worst outcome. It is scored by Traditional Chinese Medicine practitioner based on the investigators' clinical experience.
  units on a scale | 3.60 (0.77) | 3.49 (0.61) | 3.54 (0.70)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.0 (3.55) | 22.9 (2.80) | 22.9 (3.19)
Flu Vaccine [Count of Participants; unit: Participants]
  Yes | 12 | 13 | 25
  No | 58 | 55 | 113
Saliva sIgA Secretion Rate [Median (Inter-Quartile Range); unit: microgram/min] — Population: Saliva sIgA data were missing due to insufficient saliva or other procedural reasons.
  microgram/min
    number analyzed (Participants) | 47 | 45 | 92
    (all) | 93.00 [46.00 to 188.00] | 125.00 [61.00 to 211.00] | 105.5 [51.50 to 195.25]
Medication [Count of Participants; unit: Participants]
  Yes | 11 | 9 | 20
  No | 59 | 59 | 118
Supplement [Count of Participants; unit: Participants]
  Yes | 20 | 24 | 44
  No | 50 | 44 | 94
Smoking [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 70 | 67 | 137
Alcohol [Count of Participants; unit: Participants]
  Yes | 2 | 8 | 10
  No | 68 | 60 | 128

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity Score of Protective Qi Deficiency
Description: The severity score of Protective Qi Deficiency in all participants will be assessed at baseline and each follow-up visit by on-site investigators (licensed TCM practitioners). Each health condition relevant to Protective Qi Deficiency(PQD) (i.e., cold frequency, symptoms, and signs) will be scored on a designed scale (with higher number indicating more severe condition/symptom) based on a set of standardized and specified criteria (see uploaded Study Protocol for specifics). The sub-scores are then weighted (cold frequency 25%, symptoms 33.3%, signs: 41.7%) to arrive at a final PQD severity score. This score is on a 1-5 scale, with 5 being the most severe deficiency. The change of the score from baseline, indicating the treatment effect, will be calculated and analyzed by statistical means.
Time Frame: The participants PQD severity score will be re-evaluted every two weeks for a total of 12 weeks.
Population: Intent to Treat Population (all participants assigned to Proglucamune Treatment or Placebo). Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Proglucamune Treatment: Participants were treated with 2 tablets of Proglucamune per day (containing 200mg of beta glucan) for a total duration of 12 weeks.
  beta glucan: Following screening and enrollment, participants will be treated with 2 tablets (Proglucamune) per day for a total duration of 12 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).
- Placebo: Participants were treated with 2 tablets of placebo per day (contain no beta glucan) for a total duration of 12 weeks.
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
units on a scale
  PQD severity score in the Treatment group and Control group at baseline (visit 1) | 2.66 (0.45) | 2.58 (0.36)
  PQD severity score in the Treatment group and Control group at 2 weeks (visit 2) | 2.50 (0.46) | 2.57 (0.37)
  PQD severity score in the Treatment group and Control group at 4 weeks (visit 3) | 2.16 (0.60) | 2.56 (0.42)
  PQD severity score in the Treatment group and Control group at 6 weeks (visit 4) | 2.04 (0.49) | 2.48 (0.38)
  PQD severity score in the Treatment group and Control group at 8 weeks (visit 5) | 1.88 (0.50) | 2.35 (0.33)
  PQD severity score in the Treatment group and Control group at 10 weeks (visit 6) | 1.81 (0.46) | 2.30 (0.32)
  PQD severity score in the Treatment group and Control group at 12 weeks (visit 7) | 1.72 (0.43) | 2.20 (0.30)
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; It was calculated that 138 participants randomized in a 1:1 ratio between the 2 arms would have a least 90% power to detect a difference of a big effect size between Proglucamune Treatment and Placebo from baseline to week 12; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Least Square Mean Difference = -0.57, 95% CI 2-sided [-0.77 to -0.37], Standard Error of Mean 0.104

2. Primary Outcome: Change of PQD Status as Asessed by Traditional Methods.
Description: PQD status of each participant at baseline and each follow-up visit will be measured by on-site investigators (licensed TCM practitioners) through qualitative traditional assessment based on TCM practitioners' clinical experience. The status was characterized as non-PQD or PQD. The change of PQD status from baseline, indicating a treatment effect, will be calculated and analyzed by categorical statistics.
Time Frame: The participants will be followed every two weeks for a total of 12 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
Participants
  PQD status in the Treatment group and Control group at baseline (visit 1): Number of Participants Characterized as PQD | 60 | 55
  PQD status in the Treatment group and Control group at baseline (visit 1): Number of Participants Characterized as Non PQD | 10 | 13
  PQD status in the Treatment group and Control group at 2 weeks (visit 2): Number of Participants Characterized as PQD | 54 | 54
  PQD status in the Treatment group and Control group at 2 weeks (visit 2): Number of Participants Characterized as Non PQD | 16 | 14
  PQD status in the Treatment group and Control group at 4 weeks (visit 3): Number of Participants Characterized as PQD | 34 | 52
  PQD status in the Treatment group and Control group at 4 weeks (visit 3): Number of Participants Characterized as Non PQD | 36 | 16
  PQD status in the Treatment group and Control group at 6 weeks (visit 4): Number of Participants Characterized as PQD | 26 | 54
  PQD status in the Treatment group and Control group at 6 weeks (visit 4): Number of Participants Characterized as Non PQD | 44 | 14
  PQD status in the Treatment group and Control group at 8 weeks (visit 5): Number of Participants Characterized as PQD | 16 | 48
  PQD status in the Treatment group and Control group at 8 weeks (visit 5): Number of Participants Characterized as Non PQD | 54 | 20
  PQD status in the Treatment group and Control group at 10 weeks (visit 6): Number of Participants Characterized as PQD | 12 | 45
  PQD status in the Treatment group and Control group at 10 weeks (visit 6): Number of Participants Characterized as Non PQD | 58 | 23
  PQD status in the Treatment group and Control group at 12 weeks (visit 7): Number of Participants Characterized as PQD | 7 | 40
  PQD status in the Treatment group and Control group at 12 weeks (visit 7): Number of Participants Characterized as Non PQD | 63 | 28
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Chi-squared — The threshold for statistical significance was p=0.05; Risk Difference (RD) = 0.27, 95% CI 2-sided [0.10 to 0.59]

3. Secondary Outcome: Global Health_Physical Health
Description: The participants' Global Health will be assessed using the established PROMIS® Scale v1.2 . This questionnaire consists of 10 global-health related questions. The answer for nine of ten questions are graded on 1-5 scale (with 5 being the best), and one question is graded on 1 to 10 scale (with 10 being the worst grade). The sub-scores are used to obtain a final combined score of Global Health using a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores represent more. Higher scores indicate better physical health.
Time Frame: The participants will be followed every two weeks for a total of 12 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
T-score
  Physical Health Score between treatment group and control group at base line (visit 1) | 44.25 (5.66) | 44.85 (4.88)
  Physical Health Score between treatment group and control group at 2 weeks (visit 2) | 46.33 (4.97) | 45.34 (4.45)
  Physical Health Score between treatment group and control group at 4 weeks (visit 3) | 47.63 (4.85) | 45.71 (4.15)
  Physical Health Score between treatment group and control group at 6 weeks (visit 4) | 48.60 (4.98) | 46.24 (4.61)
  Physical Health Score between treatment group and control group at 8 weeks (visit 5) | 50.30 (6.22) | 46.38 (4.36)
  Physical Health Score between treatment group and control group at 10 weeks (visit 6) | 51.53 (6.52) | 46.32 (4.10)
  Physical Health Score between treatment group and control group at 12 weeks (visit 7) | 53.12 (6.82) | 47.38 (4.53)
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Least Square Mean Difference = 6.35, 95% CI 2-sided [3.93 to 8.77]

4. Secondary Outcome: Global Health_Mental Health
Description: The participants' Global Health will be assessed using the established PROMIS® Scale v1.2. This questionnaire consists of 10 global-health related questions. The answer for nine of ten questions are graded on 1-5 scale (with 5 being the best), and one question is graded on 1 to 10 scale (with 10 being the worst grade). The sub-scores are used to obtain a final combined score of Global Health using a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores present more. Higher scores indicate better mental health.
Time Frame: The participants will be followed every two weeks for a total of 12 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
T-score
  Mental Health Score between treatment group and control group at baseline (visit 1) | 45.40 (8.41) | 46.52 (6.89)
  Mental Health Score between treatment group and control group at 2 weeks (visit 2) | 46.60 (7.36) | 46.83 (6.66)
  Mental Health Score between treatment group and control group at 4 weeks (visit 3) | 48.29 (5.88) | 47.26 (6.29)
  Mental Health Score between treatment group and control group at 6 weeks (visit 4) | 48.55 (5.90) | 47.43 (6.43)
  Mental Health Score between treatment group and control group at 8 weeks (visit 5) | 49.86 (5.83) | 47.60 (6.10)
  Mental Health Score between treatment group and control group at 10 weeks (visit 6) | 50.75 (5.63) | 47.80 (5.84)
  Mental Health Score between treatment group and control group at 12 weeks (visit 7) | 51.67 (5.11) | 48.74 (5.51)
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Least Square Mean Difference = 4.049, 95% CI 2-sided [1.08 to 7.01]

5. Secondary Outcome: Saliva sIgA Secretion Rate
Description: The effect of Proglucamune on the participants' immunity will be assessed by the change of saliva secretary IgA.
Time Frame: The participants will be followed every 6 weeks during 12 week trial.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: microgram/min
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 47 | 45
microgram/min
  Saliva sIgA Secretion Rate between treatment group and control group at baseline (visit 1) | 93 [59 to 123] | 125 [79 to 145]
  Saliva sIgA Secretion Rate between treatment group and control group at 6 weeks (visit 4) | 68 [60 to 96] | 63 [51 to 86]
  Saliva sIgA Secretion Rate between treatment group and control group at 12 weeks (visit 7) | 86 [65 to 108] | 92 [70 to 109]
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; Test type: Superiority; p = 0.6, ANOVA — The threshold for statistical significance was p=0.05

6. Secondary Outcome: Emotional and Behavioral Dyscontrol - Short Form
Description: Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. This questionnaire consists of 8 questions related to emotional and behavioral control. The answers for each of the questions are graded on five levels from best to worst. A combined score is generated using a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores represent more. Higher Emotional and Behavioral Dyscontrol scores represent worse Emotional and Behavioral Dyscontrol.
Time Frame: The participants will be followed every two weeks for a total of 12 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
T-score
  Emotional&Behavioral Dyscontrol score between treatment and control groups at baseline (visit 1) | 45.80 (8.19) | 46.79 (7.93)
  Emotional&Behavioral Dyscontrol score between treatment and control groups at 2 weeks (visit 2) | 45.22 (7.65) | 45.70 (8.56)
  Emotional&Behavioral Dyscontrol score between treatment and control groups at 4 weeks (visit 3) | 45.08 (7.50) | 45.46 (8.34)
  Emotional&Behavioral Dyscontrol score between treatment and control groups at 6 weeks (visit 4) | 44.66 (7.55) | 44.42 (8.45)
  Emotional&Behavioral Dyscontrol score between treatment and control groups at 8 weeks (visit 5) | 44.25 (7.65) | 45.11 (8.11)
  Emotional&Behavioral Dyscontrol score between treatment and control groups at 10 weeks (visit 6) | 44.32 (7.78) | 44.73 (8.05)
  Emotional&Behavioral Dyscontrol score between treatment and control groups at 12 weeks (visit 7) | 38.24 (7.80) | 44.01 (7.60)
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.054, Mixed Models Analysis — The threshold for statistical significance was p=0.05

7. Secondary Outcome: Emotional Impact
Description: The participants' Emotional status will be assessed using the ASCO-Me® v2.0 Emotional Impact (Short Form). This questionnaire-based survey was established based on a Sickle-cell patient population (Please see the link http://www.ascq-me.org/Science or the citation below for detail). This questionnaire consists of 5 emotional-status related questions. The answer for each of the questions are graded on five levels from best to worst. A combined score is generated using a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores represent better health.
Time Frame: The participants will be followed every two weeks for a total of 12 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
T-score
  Emotional Impact score between treatment group and control group at baseline (visit 1) | 53.54 (6.28) | 53.43 (6.56)
  Emotional Impact score between treatment group and control group at 2 weeks (visit 2) | 54.35 (6.77) | 54.00 (7.06)
  Emotional Impact score between treatment group and control group at 4 weeks (visit 3) | 54.64 (7.17) | 53.93 (6.93)
  Emotional Impact score between treatment group and control group at 6 weeks (visit 4) | 55.11 (7.16) | 54.51 (7.13)
  Emotional Impact score between treatment group and control group at 8 weeks (visit 5) | 55.26 (7.25) | 54.34 (7.11)
  Emotional Impact score between treatment group and control group at 10 weeks (visit 6) | 56.01 (7.10) | 54.00 (7.05)
  Emotional Impact score between treatment group and control group at 12 weeks (visit 7) | 59.59 (7.07) | 55.14 (7.13)
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.13, Mixed Models Analysis — The threshold for statistical significance was p=0.05

8. Secondary Outcome: Generic Qi Change
Description: The generic Qi status of participants at baseline and each follow-up visit will be assessed by on-site investigators (licensed TCM practitioners). Each health condition relevant to generic Qi insufficiency (including history, symptoms, and signs) will be scored based on a standardized criteria, and then weighted to arrive at a final generic Qi Insufficiency Score. This score is on a 1-5 scale, with 5 being the most severe insufficiency. The change of the score from baseline, indicating the treatment effect, will be calculated and analyzed by statistical means.
Time Frame: The participants will be followed every two weeks for a total of 12 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Proglucamune Treatment | Placebo
Number analyzed (Participants) | 70 | 68
units on a scale
  Generic Qi between treatment group and control group at baseline (visit 1) | 3.09 (0.47) | 2.97 (0.40)
  Generic Qi between treatment group and control group at 2 weeks (visit 2) | 2.82 (0.48) | 2.90 (0.39)
  Generic Qi between treatment group and control group at 4 weeks (visit 3) | 2.48 (0.50) | 2.87 (0.38)
  Generic Qi between treatment group and control group at 6 weeks (visit 4) | 2.29 (0.49) | 2.83 (0.35)
  Generic Qi between treatment group and control group at 8 weeks (visit 5) | 2.14 (0.52) | 2.73 (0.34)
  Generic Qi between treatment group and control group at 10 weeks (visit 6) | 2.08 (0.48) | 2.67 (.032)
  Generic Qi between treatment group and control group at 12 weeks (visit 7) | 1.94 (0.45) | 2.58 (0.35)
Statistical Analysis 1: Comparison: Proglucamune Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Least Square Mean Difference = -0.76, 95% CI 2-sided [-0.96 to -0.56], Standard Error of Mean 0.102

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Proglucamune Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 0/70 | 0/68

LIMITATIONS AND CAVEATS:
Since the treatment (Proglucamune) is a mixture of extract from yeast and whole mushrooms (Reishi and Shiitaki), we cannot completely rule out the possibility that some compounds other than ß-glucan present in Proglucamune may have contributed to the observed effect. This is particularly so given that Reishi, known for boosting Qi in TCM, contains a variety of other biologically active compounds .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03782974/Prot_SAP_ICF_001.pdf